CLINICAL TRIAL: NCT05433116
Title: Combined Pembrolizumab and Lenvatinib After Definitive Chemoradiation of Locally Advanced HNSCC in PD-L1 Positive Patients (CPS≥1)
Brief Title: Pembrolizumab and Lenvatinib After Definitive Chemoradiation of Locally Advanced HNSCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PeLeRad; 2021-004388-28 (EudraCT Number)
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pembrolizumab + lenvatinib (Other): combined pembrolizumab (200mg q3w) and lenvatinib treatment (20mg once daily)
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib
- pembrolizumab (Other): pembrolizumab (200mg q3w)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — i.v., 200mg absolute, q3w, starting within 14 days after completion of radiochemotherapy
  Other Names: Keytruda
Drug: Lenvatinib — 20mg once daily orally, start concomitant to cycle 2 of pembrolizumab
  Other Names: Lenvima
  Arms: pembrolizumab + lenvatinib

SUMMARY:
Open-label, two-arm, prospective multicenter phase II clinical trial to determine the efficacy and safety of combined pembrolizumab and lenvatinib compared to pembrolizumab alone as maintenance therapy after definitive radiochemotherapy of locally advanced head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
This is an open-label, two-arm, prospective multicenter phase II clinical trial to determine the efficacy and safety combined pembrolizumab and lenvatinib compared to pembrolizumab alone as maintenance therapy after definitive radiochemotherapy of locally advanced head and neck squamous cell carcinoma (HNSCC). The trial will be conducted in conformance with Good Clinical Practices and subjects will be enrolled into the trial by signing the informed consent form (ICF). Only subjects with PD-L1 positive (CPS≥1) tumors according to centralized reference pathologic assessment can be enrolled. Subjects without disease progression in the study screening CT (compared to radiochemotherapy baseline CT) that fulfil all further eligibility criteria can enter the trial after completion of definitive radiochemotherapy. Sites will be required to submit tissue samples for PD-L1 assessment in central pathology.

After confirmed study inclusion, patients will be randomized to receive either combined pembrolizumab and lenvatinib (treatment arm A) or pembrolizumab alone (treatment arm B). Pembrolizumab will be administered intravenously at a dose of 200mg q3w and lenvatinib at a dose of 20mg once daily orally. The first dose of pembrolizumab has to be administered within 14 days after completion of radiochemotherapy. Treatment with lenvatinib will start concomitant to cycle 2 of pembrolizumab. Treatment will be continued until disease progression, unacceptable adverse event(s) or until the subject has received 12 months of treatment (i.e. 17 doses of pembrolizumab). Afterwards patients will enter follow-up until 24 months since study inclusion.

It is planned to randomize 48 patients. In addition, two patients are treated in advance as proof on concept with pembrolizumab and lenvatinib. Primary endpoint of the trial is the event-free survival (EFS) rate at 2 years. The aim of the trial is to increase the 2-year EFS rate from 60% to 80%. This improvement is considered to be a clinically relevant advantage.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent
2. Pathologically proven new diagnosis of squamous cell carcinoma (HNSCC) of the oral cavity, oropharynx, hypopharynx or supraglottic larynx stage III-IVB according to TMM 8th edition
3. PD-L1 combined positive score (CPS) ≥1 (in sample prior to radiochemotherapy) by central pathology review
4. Completed definitive radiochemotherapy up to at least 68Gy with at least 200mg/m² body surface area concomitant Cisplatin.
5. No progression during radiochemotherapy. Study screening CT has to be compared to radiochemotherapy baseline CT. (Study screening CT may be performed before the end of radiochemotherapy, whereas a minimum radiation dose of 50Gy has to be administered at the time point of the study screening CT.)
6. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment (pembrolizumab or lenvatinib, whichever is administered last) and refrain from donating sperm during this period. In addition, contraception has to be used for 180 days after the last dose of cisplatin.
7. Female participants:

   A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: a. Not a woman of childbearing potential (WOCBP) OR b. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment (pembrolizumab or lenvatinib, whichever is administered last). In addition, contraception has to be used for 180 days after the last dose of cisplatin.
8. The participant provides written informed consent for the trial.
9. Have measurable disease based on RECIST 1.1.
10. Have provided archival tumor tissue sample with sufficient tumor content. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
11. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
12. Have adequate organ function. Specimens must be collected within 10 days prior to the start of study intervention.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Have tumor infiltration/perforation of the skin or cervical fistula (either at timepoint of study inclusion or prior to radiochemotherapy)
2. Have radiographic evidence of major blood vessel invasion/infiltration or tumor demonstrates >90-degree abutment or encasement of a major blood vessel.
3. Had prior radical surgery for the head and neck cancer under study or induction chemotherapy with more than one cycle prior to definitive radiochemotherapy. Patients with single cycle induction chemotherapy prior radiochemotherapy can be included.
4. WOCBP who have a positive urine or serum pregnancy test within 72 hours prior to. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
5. Have received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
6. Have received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study drug administration (except from cisplatin concomitant to radiochemotherapy).
7. Have received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
8. Are currently participating in or have participated in a study of an investigational agent or have used an investigational device within 4 weeks prior to the first dose of study intervention.
9. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Have a known additional malignancy that is progressing or have required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
11. Have distant metastases.
12. Have severe hypersensitivity (≥Grade 3) to pembrolizumab, lenvatinib and/or any of their excipients.
13. Have active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
14. Have a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Have an active infection requiring systemic therapy.
16. Have a known history of Human Immunodeficiency Virus (HIV) infection.
17. Have a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
18. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment. (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of ß-hCG [or hCG]).
21. Have had an allogenic tissue/solid organ transplant.
22. Have uncontrolled blood pressure (Systolic BP>140 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.
23. Have clinically relevant electrolyte abnormalities that have not been corrected.
24. Have significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.
25. Have/had bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
26. Have > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
27. Have not recovered adequately from any toxicity from other anti- cancer treatment regimens and/or complications from major surgery prior to starting therapy. Withhold lenvatinib for at least 1 week prior to elective surgery. Do not administer for at least 2 weeks following major surgery and until adequate wound healing.
28. Have prolongation of QTc interval to >480 ms in the ECG.
29. Have a LVEF below the institutional (or local laboratory) normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO).
30. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) rate | 2 years
  To study efficacy of pembrolizumab/lenvatinib maintenance therapy versus pembrolizumab alone after definitive RCT of locally advanced HNSCC to prolong the event-free survival (EFS) rate at 2 years.

SECONDARY OUTCOMES:
Event-free survival (EFS) (continuous) | 2 years
  Pembrolizumab/lenvatinib maintenance therapy will improve further efficacy endpoints compared to expectations derived from historical data on pembrolizumab alone.
Locoregional control | Restaging 12-13 weeks after completion of radiotherapy; Follow-up every 24 weeks
  Locoregional progression will be evaluated by RECIST 1.1 criteria
Toxicity of Pembrolizumab/lenvatinib | until safety follow-up (1 year treatment + 30 days)
  Toxicity will be evaluated according to CTCAE v5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hecht, Prof., Principal Investigator — Saarland University Medical Center, Clinic for Radiotherapy and Radiooncology; Antoniu-Oreste Gostian, Prof., Study Chair — University Hospital Straubing, Clinic for Otolaryngology, Head and Neck and Facial Plastic Surgery; Henning Kahl, MD, Study Chair — University Hospital Augsburg, Radiation Oncology; Rainer Fietkau, Prof., Study Chair — University Hospital Erlangen, Radiation Oncology; Udo Gaipl, Prof., Study Chair — University Hospital Erlangen, Radiation Oncology; Markus Eckstein, MD, Study Chair — University Hospital Erlangen, Pathology
Locations (10):
- Germany (10):
  - University Hospital Ulm, Otolaryngology & Head and Neck Surgery, Ulm, Baden-Wurttemberg
  - University Hospital Augsburg, Radiation Oncology, Augsburg, Bavaria
  - University Hospital Erlangen, Radiation Oncology, Erlangen, Bavaria
  - University Hospital Regensburg, Clinic and Polyclinic for Radiotherapy, Regensburg, Bavaria
  - University Hospital Frankfurt/M, Center for Radiology, Frankfurt am Main, Hesse
  - University Hospital Giessen; Ear, nose and throat clinic, Giessen, Hesse
  - University Hospital Düsseldorf, Radiation Oncology, Düsseldorf, North Rhine-Westphalia
  - Saarland University Medical Center and Saarland University Faculty of Medicine, Clinic for Radiotherapy and Radiooncology, Homburg, Saarland
  - Hospital Chemnitz, Radiation Oncology, Chemnitz, Saxony
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden, Saxony

IPD SHARING:
Plan to Share IPD: No